CLINICAL TRIAL: NCT07031453
Title: Observational Study on the Application of Different Analgesic Regimens in Non-Mechanically Ventilated Critically Ill Patients
Brief Title: Observation and Study on the Application of Different Analgesic Regimens in Critically Ill Patients Without Mechanical Ventilation
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Li Shu, associate professor, Peking University People's Hospital
Other Study IDs: 2025-Z-40
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Patients With Moderate to Severe Pain Requiring Analgesic Medications
Keywords: Patients with moderate to severe pain requiring analgesic medications.; Sedation; respiratory depression; gastrointestinal paralysis
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Respiratory depression and gastrointestinal paralysis occurred
- No respiratory depression or gastrointestinal paralysis occurred

SUMMARY:
Pain management is a common treatment measure in the Intensive Care Unit (ICU). Due to their underlying diseases and invasive treatments, patients often experience discomfort and pain, leading to agitation, unplanned extubation, patient-ventilator asynchrony, and even neuroendocrine-immune dysregulation, sympathetic overexcitation, and impaired organ function. Analgesic therapy can reduce patient stress and increase comfort, making it an essential treatment for critically ill patients. However, it may also cause adverse effects such as respiratory depression and decreased gastrointestinal motility. There is currently no consensus on how to precisely implement analgesic therapy in non-mechanically ventilated critically ill patients to reduce adverse effects like respiratory depression.This prospective observational study will enroll non-mechanically ventilated critically ill patients receiving analgesic therapy. It will observe different analgesic strategies, including factors such as pain assessment status, drug types, duration of analgesia, and cumulative drug doses, to understand their effects and adverse reactions in non-mechanically ventilated patients. The study aims to explore optimized analgesic treatment regimens and provide evidence-based support for implementing precise analgesic therapy in clinical practice.

DETAILED DESCRIPTION:
Pain management is a critical component of treatment for critically ill patients, particularly in non-mechanically ventilated patient populations. Appropriate analgesic therapy not only impacts patient comfort but also directly influences disease outcomes and medical safety. Non-ventilated patients often endure moderate-to-severe pain due to conditions such as postoperative trauma, advanced cancer, and acute pancreatitis. Pain-induced stress responses can lead to tachycardia, hypertension, increased oxygen consumption, and immunosuppression. Studies indicate that inadequately controlled acute pain increases myocardial infarction risk by 2.3-fold and deep vein thrombosis incidence by 1.8-fold, with strong correlations to chronic pain persistence.

However, implementing analgesic therapy faces dual challenges:

1. Pain assessment tends to be delayed in patients with impaired consciousness or communication difficulties, resulting in undertreatment;
2. Analgesic drugs carry complex side-effect profiles, with opioid-associated respiratory depression occurring in 9%-12% of cases, and NSAIDs increasing gastrointestinal bleeding risk by 4.7-fold. These complications may have catastrophic consequences in non-ventilated patients. Taking respiratory depression as an example: non-ventilated patients lack artificial airway protection. Even mild reductions in respiratory rate can cause hypercapnia, potentially necessitating emergency intubation. Mortality rates among these emergently intubated patients are 3.2 times higher than those with planned intubation[3]. This therapeutic dilemma makes precise analgesic regimen selection a core clinical challenge.Notably, the novel analgesic hydromorphone-a semi-synthetic morphine derivative-exhibits 8-10 times greater analgesic potency than morphine with a non-ceiling effect. It offers rapid onset, non-toxic metabolites, and diverse administration routes, demonstrating superior clinical applicability especially in patients with hepatic/renal impairment. Preliminary studies suggest hydromorphone significantly reduces respiratory depression and gastrointestinal adverse events compared to traditional opioids. Nevertheless, clinical data in non-ventilated patients remain limited, warranting systematic evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤75 years; Non-mechanically ventilated patients (including post-extubation patients) with an anticipated ICU stay >24 hours; Patients with moderate to severe pain requiring analgesic therapy; Informed consent obtained from the patient or legal guardian.

Exclusion Criteria:

* Age <18 or >75 years; Pregnancy or lactation; Patients scheduled for general anesthesia surgery within 48 hours; Severe pre-existing parenchymal liver disease with clinically significant portal hypertension, Child-Pugh Class C cirrhosis, or acute liver failure; Bronchial asthma, COPD, or myasthenia gravis patients; Severe traumatic brain injury, brain tumors, intracranial hypertension, or other conditions predisposing to respiratory depression; History of alcohol or drug abuse; Any condition impairing cognitive assessment (e.g., language/sensory impairment or psychiatric disorders, such as aphasia or organic mental dysfunction); Inability to obtain informed consent or authorization; Participation in other investigational clinical trials within 6 months prior to screening; Known allergy to the study medication.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohort will be selected from a tertiary hospital
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The proportion of time points achieving the target analgesic score range among all time points. | The observation period starts from patient enrollment and lasts for 7 days or until transfer out of the intensive care unit (ICU).

SECONDARY OUTCOMES:
Total dosage of analgesics | The observation period starts from patient enrollment and lasts for 7 days or until transfer out of the intensive care unit (ICU).
incidence of adverse events (including but not limited to cardiovascular/respiratory depression, delayed gastrointestinal motility recovery, nausea/vomiting, and pruritus) | The observation period starts from patient enrollment and lasts for 7 days or until transfer out of the intensive care unit (ICU).
in-hospital/ICU mortality | The observation period starts from patient enrollment and lasts for 7 days or until transfer out of the intensive care unit (ICU).
length of hospital stay, and ICU length of stay | The observation period starts from patient enrollment and lasts for 7 days or until transfer out of the intensive care unit (ICU).

CONTACTS AND LOCATIONS:
Overall Officials: Shu Li, doctor, Principal Investigator — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD，all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: starting 1 year after publication
Access Criteria: The date used and/or analyzed during the current study are available from the investigator on reasonable request